CLINICAL TRIAL: NCT00735501
Title: Safety of Levemir® (Insulin Detemir) Treatment in Patients With Type 2 Diabetes
Brief Title: Observational Study to Observe the Safety of Levemir® Treatment in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1938
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency as well as dose alterations to be determined by the physician according to normal clinical evaluation
  Other Names: Levemir®

SUMMARY:
This observational study is conducted in Europe. The study aims to observe the incidence of serious adverse drug reactions in subjects with type 2 diabetes during Levemir® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with type 2 diabetes
* Currently treated with basal human insulin therapy (basal only or in combination with oral glucose lowering drugs or other insulin)
* Selection of patients will be at the discretion of the treating physician after the decision to prescribe one of the study products to the patient

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products.
* Pregnancy or breastfeeding or intention of becoming pregnant within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or above, with type 2 diabetes, who together with their physician, have decided to switch to Levemir® from human basal insulin treatment
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions, including major hypoglycaemic events | After 26 weeks

SECONDARY OUTCOMES:
Number of all hypoglycaemic events | at 12 weeks and 26 weeks
Number of all adverse drug reactions | after 12 and 26 weeks
HbA1c | at 12 and 26 weeks
Variability in fasting plasma glucose (FPG) values and average FPG levels at visits | at 12 and 26 weeks
Weight changes | at 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Copenhagen S, Denmark
- Stockholm, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com